CLINICAL TRIAL: NCT07314333
Title: A Phase 1, Single Blind, Parallel-arm Trial to Assess the Potential for Pharmacodynamic Interaction of Centanafadine When Co-administered With Stimulants in Healthy Adults
Brief Title: A Trial to Assess How Centanafadine Interacts With Stimulants in the Body
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 405-201-00198
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: ADHD
Keywords: Attention-deficit/hyperactivity disorder; Healthy Adults
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 1-(naphthalen-2-yl)-3-azabicyclo(3.1.0)hexane; Methylphenidate; Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm 1, Sequence 1: ABC (Experimental): Participants will receive dosing of centanafadine alone (A), once daily (QD) extended release (XR) capsule on Day 1 followed by methylphenidate alone (B), tablet, QD on Day 5, further followed by centanafadine, QD XR capsule along with methylphenidate, tablet (C), QD on Day 9. There will be a washout period of 96 hours between each dosing.
  Interventions: Drug: Centanafadine; Drug: Methylphenidate
- Arm 1, Sequence 2: BCA (Experimental): Participants will receive dosing of methylphenidate alone (B), tablet, QD on Day 1, followed by centanafadine, QD XR capsule along with methylphenidate, tablet (C), QD on Day 5, further followed by centanafadine alone, QD XR capsule (A) on Day 9. There will be a washout period of 96 hours between each dosing.
  Interventions: Drug: Centanafadine; Drug: Methylphenidate
- Arm 1, Sequence 3: CAB (Experimental): Participants will receive dosing of centanafadine, QD XR capsule along with methylphenidate, tablet (C), QD on Day 1, followed by centanafadine alone, QD XR capsule (A) on Day 5, further followed by methylphenidate alone, tablet (B), QD on Day 9. There will be a washout period of 96 hours between each dosing.
  Interventions: Drug: Centanafadine; Drug: Methylphenidate
- Arm 2, Sequence 1: ABC (Experimental): Participants will receive dosing of centanafadine alone, QD XR capsule (A) on Day 1 followed by lisdexamfetamine alone, capsule (B), QD on Day 5, further followed by centanafadine, QD XR capsule along with lisdexamfetamine, capsule (C), QD on Day 9. There will be a washout period of 96 hours between each dosing.
  Interventions: Drug: Centanafadine; Drug: Lisdexamfetamine
- Arm 2, Sequence 2: BCA (Experimental): Participants will receive dosing of lisdexamfetamine alone, capsule (B), QD on Day 1, followed by centanafadine, QD XR capsule along with lisdexamfetamine, capsule (C), QD on Day 5, further followed by centanafadine alone, QD XR capsule (A) on Day 9. There will be a washout period of 96 hours between each dosing.
  Interventions: Drug: Centanafadine; Drug: Lisdexamfetamine
- Arm 2, Sequence 3: CAB (Experimental): Participants will receive dosing of centanafadine, QD XR capsule along with lisdexamfetamine, capsule (C), QD on Day 1, followed by centanafadine alone, QD XR capsule (A) on Day 5, further followed by lisdexamfetamine alone, capsule (B), QD on Day 9. There will be a washout period of 96 hours between each dosing.
  Interventions: Drug: Centanafadine; Drug: Lisdexamfetamine

INTERVENTIONS:
Drug: Centanafadine — Oral, QD XR capsules.
  Other Names: EB-1020
Drug: Methylphenidate — Oral tablets.
  Other Names: Concerta
  Arms: Arm 1, Sequence 1: ABC; Arm 1, Sequence 2: BCA; Arm 1, Sequence 3: CAB
Drug: Lisdexamfetamine — Oral capsules
  Other Names: Vynase
  Arms: Arm 2, Sequence 1: ABC; Arm 2, Sequence 2: BCA; Arm 2, Sequence 3: CAB

SUMMARY:
This study will look at how centanafadine works when taken together with stimulant medicines in healthy adults, and whether combining them affects how the body responds.

DETAILED DESCRIPTION:
This is a single dose crossover study. Participants in each arm will receive 3 treatments in a 3 -sequence, 3-period, crossover design. In each arm, participants will be randomized to 1 of 3 treatment sequences: Sequence 1: ABC, Sequence 2: BCA, or Sequence 3: CAB.

Here's what each treatment incudes:

* Treatment A - centanafadine alone in both Arms 1 and 2.
* Treatment B - methylphenidate alone in Arm 1 and lisdexamfetamine alone in Arm 2.
* Treatment C - centanafadine combined with methylphenidate in Arm 1, and centanafadine combined with lisdexamfetamine in Arm 2.

The duration of trial participation for each participant will be approximately 44 days, and the overall trial duration is expected to be approximately 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.0 to 32.0 kilogram per square meter (kg/m2).
* Must be in good health, based on:

  * Medical history
  * Physical examination
  * Heart test (Electrocardiogram [ECG])
  * Lab tests (blood, urine and other routine checks)
* Willing to stay in the clinic for the required time and agree to a follow-up phone call for safety.
* Able to sign informed consent and, in the investigator's opinion, follow all trial requirements.

Exclusion Criteria:

* History of drug and/or alcohol abuse in past 2 years.
* History of or current hepatitis or acquired immune deficiency syndrome (AIDS) or carriers of hepatitis B surface antigen (HBsAg) and/or anti-hepatitis C virus (HCV), or human immunodeficiency virus (HIV) antibodies.
* Known drug allergy or hypersensitivity.
* Any history of significant bleeding problems.
* Difficulty donating blood in the past.
* Use of tobacco or exposure to second-hand smoke in the past 2 months, or high cotinine levels in blood/urine.
* Uncontrolled high blood pressure (BP) (systolic blood pressure [SBP] > 140 millimeters of mercury (mmHg) or diastolic blood pressure [DBP] > 90 mmHg) or symptomatic low blood pressure, or orthostatic hypotension (large BP drop when standing).
* History of unexplained fainting (syncope).
* Serious mental health disorders that could interfere with participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-02-05 (Actual); Primary Completion 2026-03-06 (Estimated); Study Completion 2026-03-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Blood Pressure (BP) at Day 12 or Early Termination (ET) | Baseline, Day 12 or ET
Change from Baseline in Heart Rate (HR) at Day 12 or ET | Baseline, Day 12 or ET

SECONDARY OUTCOMES:
Maximal peak plasma concentration (Cmax) for Centanafadine when co-administered with methylphenidate or lisdexamfetamine | Days 1, 5, and 9: pre-dose and at 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours post-dose
Area under the concentration time curve from time zero to the time of the last observable concentration at time (AUC0-12 hours) for Centanafadine when co-administered with methylphenidate or lisdexamfetamine | Days 1, 5, and 9: pre-dose and at 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours post-dose
Area under the concentration time curve from time zero to infinity (AUC-inf) for Centanafadine when co-administered with methylphenidate or lisdexamfetamine | Days 1, 5, and 9: pre-dose and at 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours post-dose
Time to maximum (peak) Plasma Concentration (Tmax) for Centanafadine when co-administered with methylphenidate or lisdexamfetamine | Days 1, 5, and 9: pre-dose and at 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours post-dose
Terminal phase elimination half-life (t1/2,z) for Centanafadine when co-administered with methylphenidate or lisdexamfetamine | Days 1, 5, and 9: pre-dose and at 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours post-dose
Volume of distribution following extravascular administration (Vz/F) for Centanafadine when co-administered with methylphenidate or lisdexamfetamine | Days 1, 5, and 9: pre-dose and at 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours post-dose
Apparent clearance of drug from plasma after extravascular administration (CL/F) for Centanafadine when co-administered with methylphenidate or lisdexamfetamine | Days 1, 5, and 9: pre-dose and at 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- ICON, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

REFERENCES:
- See also: Otsuka Clinical Trials Website — https://trials.otsuka-us.com/